CLINICAL TRIAL: NCT02911428
Title: Open Study of the Duration of Immunity After Vaccination With Medicinal Product GamEvac-Vector-Based Vaccine Against Ebola Virus Disease
Brief Title: Open Study of the Duration of Immunity After Vaccination With GamEvac
Status: Completed | Type: Observational
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Other Study IDs: 03 - GamEvac-2016
Record Dates: First submitted 2016-09-14; First posted 2016-09-22 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2016-09

CONDITIONS: Hemorrhagic Fever, Ebola
Keywords: Ebola; Ebola Virus Vaccines; Haemorrhagic Fever; Ebola Infection; GP protein, Ebola virus
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Hemorrhagic Fevers, Viral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The duration of immunity persistence following product administration will be assessed in healthy volunteers based on the measurements of specific antibody titers.
  * by ELISA method 12, 18 and 24 months after the vaccination vs. baseline values;
  * in virus neutralization reaction 12 months after the vaccination vs. baseline values
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- dosages of 0.25 ml: Blood sampling collection: 12, 18 and 24 months after the vaccination. The study will enroll up to 30 healthy volunteers of both genders aged 18-55 inclusive who had been earlier immunized with medicinal product GamEvac in the dosages of 0.25 ml, during the study under Protocol 02-E-2015 in October-November 2015.
  Interventions: Procedure: blood sampling collection
- dosages of 0.5 ml: Blood sampling collection: 12, 18 and 24 months after the vaccination. The study will enroll up to 30 healthy volunteers of both genders aged 18-55 inclusive who had been earlier immunized with medicinal product GamEvac in the dosages of 0.5 ml, during the study under Protocol 02-E-2015 in October-November 2015.
  Interventions: Procedure: blood sampling collection

INTERVENTIONS:
Procedure: blood sampling collection — It is an observational study; no interventions are planned in the course of common clinical practices during the study period; investigated therapeutic agents or special methods of examination will not be used in the study, except the blood sampling procedure and clinical observation specified in this Protocol.

SUMMARY:
The purpose of this study is to evaluate the post-vaccination immune status at different time points in subjects immunized against Ebola Virus Disease; to select an optimal regimen of product administration; and, to assess safety of medicinal product GamEvacVector-Based Vaccine against Ebola Virus Disease, 0.5 ml+0.5 ml/dose, following the immunization with a half (0.25 ml+0.25 ml/dose) and full (0.5 ml+0.5 ml/dose) therapeutic doses.

DETAILED DESCRIPTION:
This clinical trial is designed as an open study to evaluate the duration of immunity persistence following the administration of medicinal product GamEvac Vector-Based Vaccine against Ebola Virus Disease.

It is an observational study; no interventions are planned in the course of common clinical practices during the study period; investigated therapeutic agents or special methods of examination will not be used in the study, except the blood sampling procedure specified in this Protocol. Only those patients who have signed the information consent form for participation in the study and have been informed by physician on the objectives and methods of this project will be involved in the study.

The study consists of a single stage which is designed as a follow-up period to observe volunteers vaccinated in the course of evaluation of safety, reactogenic properties and immunogenicity of product GamEvac Vector-Based Vaccine against Ebola Virus Disease in the dosages of 0.25 ml and 0.5 ml, during the study under Protocol 02-E-2015 in October-November 2015. Vaccination will not be made within the present study. Screening of volunteers is not required: the study will involve as many of the volunteers as possible (but not more than 60 subjects) who had been immunized earlier with GamEvac Vector-Based Vaccine against Ebola Virus Disease, provided that they have no medical contraindications for blood sampling.

Study Schedule Visit 1 (outpatient): the goal of this visit is to assess whether a patient meets the inclusion/exclusion criteria. All procedures should be carried out upon receipt of the informed consent form signed by patient. The visit will be held 12 months after the vaccination.

Visit 2 (outpatient): 18 months after the vaccination. Visit 3 (outpatient): 24 months after the vaccination. The duration of immunity persistence following product administration will be assessed in healthy volunteers based on the measurements of specific antibody titers.

by ELISA method 12, 18 and 24 months after the vaccination vs. baseline values; in virus neutralization reaction 12 months after the vaccination vs. baseline values.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-56 who had been earlier vaccinated with medicinal product GamEvac in the dosages of 0.25 ml and 0.5 ml, during the study under Protocol 02-E-2015 in October-November 2015.
* Written informed consent signed by patients prior to their involvement in the study

Exclusion Criteria:

* Absence of the earlier vaccination with medicinal product GamEvac in the dosages of 0.25 ml and 0.5 ml, during the study under Protocol 02-E-2015 in October-November 2015.
* Presence of a concomitant illness which could preclude obtaining a venous blood sample or affect the study process: (critical patient's condition, seizures, agitated state, blood loss and shocks of different origin).

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will enroll up to 60 healthy volunteers of both genders aged 18-55 inclusive who had been earlier immunized with medicinal product GamEvac in the dosages of 0.25 ml and 0.5 ml, during the study under Protocol 02-E-2015 in October-November 2015.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2017-12-25 (Actual); Study Completion 2017-12-25 (Actual)

PRIMARY OUTCOMES:
duration of immunity using ELISA method | 12 months after the vaccination
  To evaluate the duration of immunity persistence following the product administration in healthy volunteers by measuring the specific antibody titer:
  - using ELISA method 12 months after the vaccination vs. baseline values
duration of immunity using ELISA method | 18 months after the vaccination
  To evaluate the duration of immunity persistence following the product administration in healthy volunteers by measuring the specific antibody titer:
  - using ELISA method 18 months after the vaccination vs. baseline values
duration of immunity using ELISA method | 24 months after the vaccination
  To evaluate the duration of immunity persistence following the product administration in healthy volunteers by measuring the specific antibody titer:
  - using ELISA method 24 months after the vaccination vs. baseline values

SECONDARY OUTCOMES:
duration of immunity in virus neutralization reaction | 12 months after the vaccination vs. baseline values
  To evaluate the duration of immunity persistence following the product administration in healthy volunteers by measuring the specific antibody titer
Incidence of Treatment-Emergent Adverse Events | 12, 18 and 24 months after the vaccination
  Incidence of Treatment-Emergent Adverse Events. To assess product safety by collecting information on adverse events, development of infectious and non-infectious diseases, and on cases where vaccinated volunteers were seeking for medical care during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin Zhdanov, MD, PhD, Principal Investigator — Federal state budget military educational institution of higher education "Military medical Academy named after S. M. Kirov" Ministry of defense of the Russian Federation
Locations (1):
- Federal state budget military educational institution of higher education "Military medical Academy named after S. M. Kirov" Ministry of defense of the Russian Federation, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided